CLINICAL TRIAL: NCT03124914
Title: Relationship Between Neuromuscular Fatigue, Perceived Tiredness and Level Of Physical Activity of Patients Living With HIV
Acronym: ACT PHY HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-PP-05
Record Dates: First submitted 2016-12-30; First posted 2017-04-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: HIV Seropositivity
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients considered physically active (Active Comparator): Measures of strength and determination of neuromuscular fatigue
  Interventions: Other: Neuromuscular tests
- Patients considered physically inactive (Active Comparator): Measures of strength and determination of neuromuscular fatigue
  Interventions: Other: Neuromuscular tests

INTERVENTIONS:
Other: Neuromuscular tests — Neuromuscular tests

SUMMARY:
Fatigue is a common symptom in people living with HIV (PHAs) that affects all aspects of life . This would include physical deconditioning, a reduction in motor skills . Numerous studies show that physical activity brings benefits for the quality of life of PHAs . However, due to the predominantly reported fatigue, many PHAs are not physically active enough in relation to these recommendations. While it is recognized that fatigue is predominant in PHAs, this complaint has mainly been subjectively quantified and has rarely been physically objectified a better understanding of the relationship between neuromuscular fatigue, perceived fatigue and the level of physical activity of PHAs is needed in line with current work on integrating fatigue.

OBJECTIVES This project, based on an integrative (eg, neurophysiological and psychological) approach to fatigue, aims to better explain and prevent the vicious circle of physical deconditioning in PHAs by examining the relationships between neuromuscular fatigue, perceived fatigue, Physical activity of patients.

The main objective of the study will be to compare the characteristics of neuromuscular fatigue in physically active or inactive PHAs.

The secondary objective will be to examine the relationship between neuromuscular fatigue, level of physical activity and perceived physical fatigue of PHAs.

CONDUCT OF THE STUDY Cross-sectional comparative study without individual benefit for the patient. Monocentric test to quantify and relate neuromuscular fatigue, perceived physical fatigue, and physical activity level. The main inclusion criteria for this study are: PLHIV aged between 40 and 60; Diagnosed and treated with antivirals after 1996, irrespective of the value of the viral load and CD4 lymphocyte level at the last assessment; The physical activity level of the patients will be evaluated before the start of the study in order to constitute two distinct groups

* Principal evaluation criterion: Investigation of the neurophysiological characteristics of fatigue will be done by recording the capacity to produce force at the level of the extensor muscles of the knee under conditions of voluntary contractions and evoked by magnetic stimulation at the level of Femoral nerve.
* Secondary evaluation criteria: the investigation of the perceived fatigue will be done by a valid psychometric questionnaire.

DETAILED DESCRIPTION:
RATIONAL Fatigue is a common symptom in people living with HIV (PHAs) that affects all aspects of life . This would include physical deconditioning, a reduction in motor skills . Numerous studies show that physical activity brings benefits for the quality of life of PHAs. However, due to the predominantly reported fatigue, many PHAs are not physically active enough in relation to these recommendations. While it is recognized that fatigue is predominant in PHAs, this complaint has mainly been subjectively quantified and has rarely been physically objectified. , a better understanding of the relationship between neuromuscular fatigue, perceived fatigue and the level of physical activity of PHAs is needed in line with current work on integrating fatigue.

OBJECTIVES OF THE STUDY This project, based on an integrative (eg, neurophysiological and psychological) approach to fatigue, aims to better explain and prevent the vicious circle of physical deconditioning in PHAs by examining the relationships between neuromuscular fatigue, perceived fatigue, Physical activity of patients.

The main objective of the study will be to compare the characteristics of neuromuscular fatigue in physically active or inactive PHAs.

The secondary objective will be to examine the relationship between neuromuscular fatigue, level of physical activity and perceived physical fatigue of PHAs.

CONDUCT OF THE STUDY Cross-sectional comparative study without individual benefit for the patient. Monocentric test to quantify and relate neuromuscular fatigue, perceived physical fatigue, and physical activity level. The main inclusion criteria for this study are: PLHIV aged between 40 and 60; Diagnosed and treated with antivirals after 1996, irrespective of the value of the viral load and CD4 lymphocyte level at the last assessment; The physical activity level of the patients will be evaluated before the start of the study in order to constitute two distinct groups: (a) a group of patients considered as physically active (SAP> 22) and (b) a group of patients considered as Physically inactive (SAP <15). Confirmed by blood diagnosis. Those who have recently stopped their antiretroviral treatment and / or their medical follow-up and who have a progressive recovery of their infection and those affected by other health conditions marked by fatigue will be excluded.

* Principal evaluation criterion: Investigation of the neurophysiological characteristics of fatigue will be done by recording the capacity to produce force at the level of the extensor muscles of the knee under conditions of voluntary contractions and evoked by magnetic stimulation at the level of Femoral nerve.
* Secondary evaluation criteria: the investigation of the perceived fatigue will be done by a valid psychometric questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* HIV patient - PLHIV (person living with HIV)
* Patient aged between 40 and 60
* patient attended the Nice University Hospital

Exclusion Criteria:

* Patient refusing to sign informed consent
* Subjects with motor disabilities;
* Subjects incapable of answering questionnaires independently;
* Subjects with anosognosia;
* Subjects with contraindications to physical practice;
* Persons co-infected with HCV or HBV
* People with associated fatigue-associated comorbidity (renal disease, cancer, multiple sclerosis (Harmon et al., 2008)
* Women who have been pregnant or have given birth in the previous twelve months
* Subjects with contraindications to magnetic stimulation (hearing disorders or carriers of metallic material.
* Subjects under tutelage, under curatorship or under safeguard of justice;
* Persons deprived of their liberty (administrative or judicial).
* Persons hospitalized without consent
* Persons admitted to a health or social institution for purposes other than research
* Persons of legal age who are the object of a legal protection measure or who are unable to express their consent

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
relationship between neuromuscular fatigue, perceived fatigue and the level of physical activity | through study completion, 1 year after the start

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No